CLINICAL TRIAL: NCT00041197
Title: A Phase III Randomized Double-Blind Study of Adjuvant STI571 (Gleevec™) Versus Placebo in Patients Following the Resection of Primary Gastrointestinal Stromal Tumor (GIST)
Brief Title: Imatinib Mesylate in Treating Patients With Primary Gastrointestinal Stromal Tumor That Has Been Completely Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02930; Z9001; CDR0000069452; U10CA076001 (NIH)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate (Gleevec; STI571) once daily. Treatment continues for 1 year in the absence of unacceptable toxicity. Patients who develop a recurrence during the year of initial treatment receive imatinib mesylate (Gleevec; STI571) at an increased dose. Patients who develop a recurrence after the year of initial treatment restart imatinib mesylate (Gleevec; STI571) and continue taking the drug at the discretion of the principal investigator.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis
- Arm II (placebo) (Placebo Comparator): Patients receive oral placebo once daily. Treatment continues for 1 year in the absence of unacceptable toxicity. Patients who develop a recurrence at any time discontinue placebo and crossover to arm I. Treatment on arm I continues at the discretion of the principal investigator.
  Interventions: Other: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given orally (PO)
  Other Names: CGP 57148; Gleevec; Glivec
  Arms: Arm I (imatinib mesylate)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase III trial is studying imatinib mesylate to see how well it works compared to placebo in treating patients with primary gastrointestinal stromal tumor that has been completely removed by surgery. Imatinib mesylate may interfere with the growth of tumor cells and may be an effective treatment for patients with primary gastrointestinal stromal tumor that has been completely removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether patients with resected primary gastrointestinal stromal tumor (GIST) who are randomized to the STI571 (imatinib mesylate) Arm have longer recurrence-free survival as compared to the patients randomized to the placebo Arm.

SECONDARY OBJECTIVES:

I. To ascertain whether patients with resected primary GIST who are randomized to the STI571 Arm have longer survival as compared to the patients randomized to the placebo Arm.

II. To obtain from patients with GIST: tumor tissue (before therapy with STI571 and if the patient develops recurrence), blood specimens (before therapy with STI571), and serum specimens (before therapy with STI571, after completing therapy with STI571, and if the patient develops recurrence) for scientific correlative analyses.

III. To assess the safety/efficacy of oral STI571 therapy in the adjuvant setting.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral imatinib mesylate (Gleevec; STI571) once daily. Treatment continues for 1 year in the absence of unacceptable toxicity. Patients who develop a recurrence during the year of initial treatment receive imatinib mesylate (Gleevec; STI571) at an increased dose. Patients who develop a recurrence after the year of initial treatment restart imatinib mesylate (Gleevec; STI571) and continue taking the drug at the discretion of the principal investigator.

ARM II: Patients receive oral placebo once daily. Treatment continues for 1 year in the absence of unacceptable toxicity. Patients who develop a recurrence at any time discontinue placebo and crossover to arm I. Treatment on arm I continues at the discretion of the principal investigator.

Patients are followed every 3 months for 2 years, then every 6 months for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have an ECOG/Zubrod performance status of =< 2
* Patient must have a histologic diagnosis of primary GIST (without peritoneal or distant metastasis) that expresses Kit protein by immunohistochemistry and have tumor size >= 3cm in maximum dimension
* Patient must have undergone complete gross resection (includes R0 [negative microscopic margins] and R1 [positive microscopic margins]) of a primary GIST within 70 days prior to registration
* Patient must have a chest x-ray completed within 28 days prior to registration; NOTE: Chest CT within 28 days prior to registration can be used in lieu of chest x-ray
* Patient must have a post-operative CT scan with IV and PO contrast or MRI with contrast (if allergic to CT contrast) of abdomen and pelvis within 28 days prior to registration
* Creatinine =< 1.5 times the institution ULN
* WBC >= 2,000/mm^3
* Platelets >= 100,000/mm^3
* Total Bilirubin =< 1.5 times the institution ULN; NOTE: Patients with elevated bilirubin secondary to Gilbert's disease are eligible to participate in the study
* AST =< 2.5 times the institution ULN
* ALT =< 2.5 times the institution ULN
* Female of childbearing potential must have negative serum pregnancy test; NOTE: Post-menopausal women must be amenorrheic for at least 12 months to be deemed not of reproductive potential
* Patient or the patient's legally acceptable representative must provide a signed and dated written informed consent prior to registration and any study-related procedures
* Patient must provide written authorization to allow the use and disclosure of their protected health information; NOTE: This may be obtained in either the study-specific informed consent or in a separate authorization form and must be obtained from the patient prior to study registration (non-US sites are exempt from HIPAA regulations)
* If patient is a cancer survivor, ALL of the following criteria apply:

  * Patient has undergone potentially curative therapy for all prior malignancies
  * No evidence of any prior malignancies for at least 5 years with no evidence of recurrence (except for effectively treated basal cell or squamous carcinoma of the skin, carcinoma in-situ of the cervix that has been effectively treated by surgery alone, or lobular carcinoma in-situ of the ipsilateral or contralateral breast treated by surgery alone)
  * Patient is deemed by their treating physician to be at low risk for recurrence from prior malignancies

Exclusion Criteria:

* Patient has received post-operative chemotherapy
* Patient has received post-operative radiation therapy
* Patient has received post-operative investigational treatment
* Patient has received prior therapy with STI571
* Patient has had an active infection requiring antibiotics within 14 days prior to registration
* Patient has objective evidence of residual disease on the postoperative CT scan or MRI of the abdomen or pelvis
* Patient, if female and breastfeeding; NOTE: It is not known whether STI571or its metabolites are excreted in human milk; however, in lactating female rats administered 100mg/kg, a dose approximately equal to the maximum clinical dose of 800mg/day based on body surface area, STI571 and /or its metabolites were extensively excreted in milk; it is estimated that approximately 1.5% of a maternal dose is excreted into milk, which is equivalent to a dose to the infant of 30% the maternal dose per unit body weight; women should be advised against breastfeeding while taking STI571
* Patient has New York Heart Association class 3 or 4 cardiac disease
* Patient is taking full dose warfarin; NOTE: The use of mini-dose warfarin (1mg orally per day) for prevention of central line-associated deep venous thrombosis is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Actual)
Dates: Start 2002-06; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | From date of resection to the date of first observation of recurrence, assessed up to 10 years
  An O'Brien-Fleming bound will be used to stop the trial early for superiority of the STI571 arm.

SECONDARY OUTCOMES:
Safety as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 5 years
  Safety analysis will consist of routine tabulations, detailed documentation concerning all adverse events, detailed documentation of any unusual events, and any special reports, analyses, or tabulations requested by the DSMC.
Relationship between genetic and phenotypic characteristics of GIST and clinical outcomes | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald DeMatteo, Principal Investigator — American College of Surgeons
Locations (1):
- American College of Surgeons Oncology Group, Durham, North Carolina, United States

REFERENCES:
- [Derived] Corless CL, Ballman KV, Antonescu CR, Kolesnikova V, Maki RG, Pisters PW, Blackstein ME, Blanke CD, Demetri GD, Heinrich MC, von Mehren M, Patel S, McCarter MD, Owzar K, DeMatteo RP. Pathologic and molecular features correlate with long-term outcome after adjuvant therapy of resected primary GI stromal tumor: the ACOSOG Z9001 trial. J Clin Oncol. 2014 May 20;32(15):1563-70. doi: 10.1200/JCO.2013.51.2046. Epub 2014 Mar 17. PMID 24638003
- [Derived] Dematteo RP, Ballman KV, Antonescu CR, Maki RG, Pisters PW, Demetri GD, Blackstein ME, Blanke CD, von Mehren M, Brennan MF, Patel S, McCarter MD, Polikoff JA, Tan BR, Owzar K; American College of Surgeons Oncology Group (ACOSOG) Intergroup Adjuvant GIST Study Team. Adjuvant imatinib mesylate after resection of localised, primary gastrointestinal stromal tumour: a randomised, double-blind, placebo-controlled trial. Lancet. 2009 Mar 28;373(9669):1097-104. doi: 10.1016/S0140-6736(09)60500-6. Epub 2009 Mar 18. PMID 19303137